CLINICAL TRIAL: NCT06415032
Title: Comparison of 'Quilting Sutures' With 'Conventional Sutures and Drain Placement' After Mastectomy: a Multicentre, Pragmatic Randomised Controlled Trial
Brief Title: Quilting Sutures After Mastectomy
Acronym: BE-Quilt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S66948
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: Mastectomy; Drain policy; Pain; Upper limb function; Cosmetic outcome; Quilting
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Mastectomy

STUDY DESIGN:
Intervention Model Description: A multicentre, pragmatic randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quilting sutures without drain placement (Experimental)
  Interventions: Procedure: Mastectomy with Quilting sutures without drain placement
- Conventional sutures with drain placement (Active Comparator)
  Interventions: Procedure: Mastectomy with Conventional sutures with drain placement

INTERVENTIONS:
Procedure: Mastectomy with Quilting sutures without drain placement — The nipple-areola complex is removed, and dissection of skin flaps is performed using electrocautery. The breast tissue, including the prepectoral fascia is removed from the pectoral muscle. After the mastectomy, the skin flaps are sutured onto the pectoral muscle using polyfilament absorbable sutures (e.g. Stratafix PDS® 1 CT needle) placed at 4- to 5-cm intervals in two or three rows depending on the extent of the skin flaps. Care is taken to prevent dimpling of the skin. The axillary region is also approximated. Care is taken to prevent damage to nerves and blood vessels. No suction drains are placed. For skin closure, the edges are sutured using absorbable monofilament sutures (e.g. Biosyn l® 3-0, Monocryl® 3-0) depending on the surgeon's preference.
  Arms: Quilting sutures without drain placement
Procedure: Mastectomy with Conventional sutures with drain placement — The nipple-areola complex is removed, and dissection of skin flaps is performed using electrocautery. The breast tissue, including the prepectoral fascia is removed from the pectoral muscle. After mastectomy no flap fixation is performed. The skin is closed in a conventional manner using an absorbable skin suture. One or two suction drains are placed before skin closure. The drains are placed in the mastectomy gutter lateral to the pectoral muscle and/or in the prepectoral area. For skin closure, the edges are sutured using absorbable monofilament sutures (e.g. Biosyn l® 3-0, Monocryl® 3-0) depending on the surgeon's preference. Drain output is recorded daily. Drain removal policy varies among participating centres. In some centres drain removal is based on volume of drained fluids while in other centres it depends on the postoperative time
  Arms: Conventional sutures with drain placement

SUMMARY:
The use of wound drains after mastectomy is common practice in Belgium. However, placement of suction drainage has several disadvantages. Skin bacteria can enter via the drain and cause infection, or the drain itself can cause discomfort and a need for daily nursing. After drain removal, seroma is the most common complication following breast cancer surgery. Seromas are collections of serous fluid that frequently develop under the skin or in the axillary space formed after mastectomy and/or axillary lymph node dissection, resulting from surgical trauma to blood/lymphatic vessels and post-traumatic inflammation. Seroma formation can cause discomfort and limitations in shoulder function. Moreover, it is associated with surgical site infections, often requires treatment and increases healthcare consumption. Wound healing problems might be a cause of postponement of adjuvant therapy.

The quilting suture technique, in which the skin is sutured to the pectoralis muscle and drain placement is not needed, may lead to a significant reduction of seroma with a decrease in the number of aspirations and surgical site infections.

In this national multicentric study, we will compare mastectomy with placement of suction drains, a standard technique used in the vast majority of Belgian hospitals, with the new quilting suture technique without placement of suction drains. We will focus on 3 distinct primary outcomes:

* Pain of the mastectomy area 6 months after surgery
* Upper limb function 6 months after surgery
* Cosmetic outcome scored by the patient 6 months after surgery.

The goal of this study is to demonstrate the absence of long-term negative effects of the quilting suture technique on shoulder function, cosmetic outcome, and pain management.

ELIGIBILITY:
Inclusion Criteria:

* capable of giving written informed consent
* age ≥ 18 years
* scheduled for unilateral mastectomy without immediate breast reconstruction with or without axillary surgery (sentinel lymph node biopsy or axillary lymph node dissection)

Exclusion Criteria:

* scheduled for mastectomy with immediate breast reconstruction
* scheduled for synchronous bilateral breast and/or axillary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Pain in the mastectomy area scored by VAS | 6 months postoperative
  A non-inferiority margin of 10 mm was adopted, which implies that a difference between both arms up to 10 mm in favour of the standard approach would be clinically acceptable
Upper limb function scored by QuickDASH | 6 months postoperative
  A non-inferiority margin of 10 points was adopted, which implies that a difference between both arms up to 10 points in favour of the standard approach would be clinically acceptable.
Cosmetic outcome scored by the patient on a 10-point scale | 6 months postoperative
  A non-inferiority margin of 1 point on the 10-point scale was adopted which implies that a difference between both arms up to 1 point in favour of the standard approach would be clinically acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Ann Smeets, MD,PhD, Principal Investigator — UZ Leuven
Locations (1):
- Surgical Oncology, UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No